CLINICAL TRIAL: NCT05612074
Title: Kinetics of Methemoglobin Concentration in Healthy Subjects Exposed to High Dose Inhaled Nitric Oxide
Brief Title: Methemoglobin Concentration in High Dose Inhaled Nitric Oxide
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Medical Director, Respiratory Care, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022P002884
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
Keywords: nitric oxide; methemoglobin; nitrogen dioxide
MeSH Terms: interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Physiologic study in healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nitric Oxide (Experimental): High dose inhaled nitric oxide (targeting 250 ppm and not exceeding 300 ppm) in a nitrogen-oxygen-air mixture, at two different FiO2 levels (0.21 and 0.8) will be delivered intermittently with a dedicated system and a snug-fitting facemask to healthy volunteers three times per day for 5 days. The subjects will be monitored before, during and after the administration
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhaled nitric oxide (Medical grade, in NO/N2 tanks) will be delivered in a oxygen-air-nitrogen mixture for 30 minutes three times per day
  Other Names: Nitric Oxide; Gaseous Nitric Oxide

SUMMARY:
The goal of this clinical trial is to learn about the kinetic of methemoglobin in healthy subjects breathing high dose inhaled nitric oxide.

The main questions it aims to answer are:

* What are the kinetics of methemoglobin formation at a maximum of 300 parts per million of nitric oxide and oxygen
* What are the kinetics of methemoglobin reduction after nitric oxide discontinuation

Participants will be exposed to intermittent high dose inhaled nitric oxide at a maximum of 300 parts per million while being continuously monitored.

DETAILED DESCRIPTION:
The current proposed physiologic study is a single center, open-label clinical trial in healthy subjects. The primary aim is to describe kinetics of methemoglobin (MetHb) formation and reduction during exposure to high dose inhaled nitric oxide (iNO) at a maximum of 300 parts per million in healthy volunteers. The investigators will also assess the contribution of increased cardiac output in relation to MetHb formation/reduction and of different inspired oxygen concentrations on the production of nitrogen dioxide (NO2).

The study protocol consists of breathing iNO at a maximum of 300 parts per million (ppm) and two different FiO2 levels (i.e. 21% and 80%). The combination of iNO and FiO2 levels identifies 2 study cohorts; five different subjects will be enrolled for each cohort. The maximum number of volunteers enrolled in this clinical trial is 10 spontaneously breathing, awake, healthy subjects, divided in two groups (5 volunteers/group, 2 groups). The first 5 subjects will be exposed to iNO in a mixture of gas at 21% of FiO2, the second group of 5 patients will receive iNO a mixture of gas at 80% of FiO2. Each volunteer will be exposed to a maximum of 300 ppm of iNO at 3 times/day for 5 consecutive days. Thus, a maximum of 150 total iNO treatments will be administered (10 enrolled volunteers, 5 days, 3 treatments/day). On the fifth day of the study, the iNO administration will be performed during physical exercise that will increase the respiratory rate of the subject, in order to study the influence of the respiratory rate on the rate of MetHb formation. During each treatment period, a threshold of MetHb = 10% and/or inspiratory NO2 = 5 ppm (as defined by the OSHA, https://www.osha.gov/chemicaldata/21, last accessed on Oct 31, 2022) will be used as stopping criteria for gas inhalation. Also, iNO administration will be stopped at any time, regardless of the MetHb and NO2 levels, at the discretion of the subject.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 64 years-old volunteers.
* Body Mass Index (BMI) 18 - 30 kg/m2.
* Absence of current systemic and/or respiratory diseases.
* Capacity to consent to the study.

Exclusion Criteria:

* Evidence of any physical, mental, and/or medical conditions that would make the proposed studies relatively more hazardous.
* Systemic and/or respiratory disease with or without any functional limitation.
* Left ventricle ejection fraction < 30%.
* Baseline MetHb ≥ 3%
* Other conditions of increased risk for MetHb formation: genetic diseases (e.g., glucose-6-phosphate dehydrogenase deficiency, cytochrome b5 reductase deficiency, sickle cell disease), significant anemia or baseline elevation in MetHb.
* History of transient ischemic attack or stroke.
* Active smoking and tobacco chewers. Volunteers may be enrolled if they quit smoking for more than 1 year and less than 10 pack years total.
* Any vaping/e-cigarettes use
* Excess alcohol use: more than ½ L/day of wine consumption or equivalent
* Current use of any recreational drugs (including the use of medical marijuana) or use of recreational drugs over the past year.
* Pregnancy determined by blood pregnancy test detecting presence of human chorionic gonadotropin (hCG).
* Less than six weeks postpartum.
* Any current medication uses except oral contraceptives.
* Lower respiratory infection within the last 30 days.
* Claustrophobia (inability to wear a facemask) or other active psychiatric conditions or unwillingness to cooperate with the investigators and other medical teams.
* Currently enrolled in another research study.
* Facial abnormalities that would preclude proper use of a face mask.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Methemoglobin kinetics | 7 days
  Levels of methemoglobin formation and reduction during and after exposure to high dose inhaled nitric oxide

SECONDARY OUTCOMES:
Nitric Oxide Metabolites | 7 days
  Measurement of Nitric Oxide metabolites (urinary and plasma) in subjects exposed to high dose iNO.
Nitrogen Dioxide | 5 days
  Inspiratory NO2 concentrations at different inspiratory concentrations of NO and O2

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiegand SB, Traeger L, Nguyen HK, Rouillard KR, Fischbach A, Zadek F, Ichinose F, Schoenfisch MH, Carroll RW, Bloch DB, Zapol WM. Antimicrobial effects of nitric oxide in murine models of Klebsiella pneumonia. Redox Biol. 2021 Feb;39:101826. doi: 10.1016/j.redox.2020.101826. Epub 2020 Dec 11. PMID 33352464
- [Background] Di Fenza R, Yu B, Carroll RW, Berra L. Chemiluminescence-based Assays for Detection of Nitric Oxide and its Derivatives from Autoxidation and Nitrosated Compounds. J Vis Exp. 2022 Feb 16;(180). doi: 10.3791/63107. PMID 35253799
- [Background] Valsecchi C, Winterton D, Safaee Fakhr B, Collier AY, Nozari A, Ortoleva J, Mukerji S, Gibson LE, Carroll RW, Shaefi S, Pinciroli R, La Vita C, Ackman JB, Hohmann E, Arora P, Barth WH Jr, Kaimal A, Ichinose F, Berra L; DELiverly oF iNO (DELFiNO) Network Collaborators. High-Dose Inhaled Nitric Oxide for the Treatment of Spontaneously Breathing Pregnant Patients With Severe Coronavirus Disease 2019 (COVID-19) Pneumonia. Obstet Gynecol. 2022 Aug 1;140(2):195-203. doi: 10.1097/AOG.0000000000004847. Epub 2022 Jul 6. PMID 35852269
- [Background] Safaee Fakhr B, Di Fenza R, Gianni S, Wiegand SB, Miyazaki Y, Araujo Morais CC, Gibson LE, Chang MG, Mueller AL, Rodriguez-Lopez JM, Ackman JB, Arora P, Scott LK, Bloch DB, Zapol WM, Carroll RW, Ichinose F, Berra L; Nitric Oxide Study Investigators. Inhaled high dose nitric oxide is a safe and effective respiratory treatment in spontaneous breathing hospitalized patients with COVID-19 pneumonia. Nitric Oxide. 2021 Nov 1;116:7-13. doi: 10.1016/j.niox.2021.08.003. Epub 2021 Aug 13. PMID 34400339
- [Background] Bartley BL, Gardner KJ, Spina S, Hurley BP, Campeau D, Berra L, Yonker LM, Carroll RW. High-Dose Inhaled Nitric Oxide as Adjunct Therapy in Cystic Fibrosis Targeting Burkholderia multivorans. Case Rep Pediatr. 2020 Jun 24;2020:1536714. doi: 10.1155/2020/1536714. eCollection 2020. PMID 32685229
- [Background] Miller C, Miller M, McMullin B, Regev G, Serghides L, Kain K, Road J, Av-Gay Y. A phase I clinical study of inhaled nitric oxide in healthy adults. J Cyst Fibros. 2012 Jul;11(4):324-31. doi: 10.1016/j.jcf.2012.01.003. Epub 2012 Apr 18. PMID 22520076
- [Background] Wiegand SB, Safaee Fakhr B, Carroll RW, Zapol WM, Kacmarek RM, Berra L. Rescue Treatment With High-Dose Gaseous Nitric Oxide in Spontaneously Breathing Patients With Severe Coronavirus Disease 2019. Crit Care Explor. 2020 Nov 16;2(11):e0277. doi: 10.1097/CCE.0000000000000277. eCollection 2020 Nov. PMID 33225304
- [Background] Safaee Fakhr B, Wiegand SB, Pinciroli R, Gianni S, Morais CCA, Ikeda T, Miyazaki Y, Marutani E, Di Fenza R, Larson GM, Parcha V, Gibson LE, Chang MG, Arora P, Carroll RW, Kacmarek RM, Ichinose F, Barth WH Jr, Kaimal A, Hohmann EL, Zapol WM, Berra L. High Concentrations of Nitric Oxide Inhalation Therapy in Pregnant Patients With Severe Coronavirus Disease 2019 (COVID-19). Obstet Gynecol. 2020 Dec;136(6):1109-1113. doi: 10.1097/AOG.0000000000004128. PMID 32852324
- [Background] Pinciroli R, Traeger L, Fischbach A, Gianni S, Morais CCA, Fakhr BS, Di Fenza R, Robinson D, Carroll R, Zapol WM, Berra L. A Novel Inhalation Mask System to Deliver High Concentrations of Nitric Oxide Gas in Spontaneously Breathing Subjects. J Vis Exp. 2021 May 4;(171). doi: 10.3791/61769. PMID 34028428
- [Background] Gianni S, Fenza RD, Morais CCA, Fakhr BS, Mueller AL, Yu B, Carroll RW, Ichinose F, Zapol WM, Berra L. High-Dose Nitric Oxide From Pressurized Cylinders and Nitric Oxide Produced by an Electric Generator From Air. Respir Care. 2022 Feb;67(2):201-208. doi: 10.4187/respcare.09308. Epub 2021 Aug 19. PMID 34413210